CLINICAL TRIAL: NCT00200148
Title: A Prospective Randomized Trial of Acute Normovolemic Hemodilution Compared to Standard Intraoperative Management in Patients Undergoing Major Hepatic Resection and Pancreaticoduodenectomy
Brief Title: Acute Normovolemic Hemodilution Versus Standard Intraoperative Management in Patients Having Hepatic Resection and Pancreaticoduodenectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 04-004
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Pancreaticoduodenectomy; Hepatectomy
Keywords: Pancreaticoduodenectomy; Hepatectomy; Major Hepatic resection; Acute Normovolemic Hemodilution
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- 1 (Experimental): For patients randomized to ANH
  Interventions: Procedure: Normovolemic Hemodilution (ANH)
- 2 (Active Comparator): standard intraoperative management
  Interventions: Procedure: Standard of care

INTERVENTIONS:
Procedure: Normovolemic Hemodilution (ANH) — For those patients randomized to ANH, the pre-calculated volume of blood will be withdrawn to a target hemoglobin of 8.0 - 8.5 g/dl (maximum of 3 L) using the formula VL=EBV x (HO-HF)/Hav, as above. The removed blood will be stored in a standard citrate-phosphate-dextrose buffer solution in blood storage bags in the operating room. During removal of blood, colloid and crystalloid solutions will be administered via peripheral intravenous lines in order to maintain euvolemia. For all patients, arterial blood will be sampled every 30 minutes during the resection for assessment of arterial blood gases/pH; Hgb levels will be measured every 30 minutes.For patients randomized to ANH, autologous blood will be re-infused in the reverse order from which it was removed, and allogeneic blood will given only after all autologous blood has been given.
  Arms: 1
Procedure: Standard of care — An 8.5 French central venous catheter and an arterial line will be placed in all patients. If the patient has a central line already in place, this may be used in place of the 8.5 French internal jugular catheter. Continuous monitoring of heart rate, blood pressure, ECG (II, V5), CVP, end tidal CO2, oxygen saturation, temperature and urine output will be performed for all patients.For all hepatic resections, standard low CVP anesthetic management will be employed.For all patients, arterial blood will be sampled every 30 minutes during the resection for assessment of arterial blood gases/pH; Hgb levels will be measured every 30 minutes.All patients will receive standard postoperative management. Routine laboratory studies, including comprehensive panel, CBC and coagulation profile, will be obtained daily in the post-operative period.
  Arms: 2

SUMMARY:
With a major liver or pancreas operation, there is a chance that one will require a transfusion of blood products (either red blood cells or plasma). This may be necessary during the operation or a few days after surgery. The surgeons at Memorial Sloan-Kettering Cancer Center perform a very large number of liver or pancreas resections every year and have pioneered techniques that minimize bleeding during the operation. Even so, liver or pancreas operations such as the one that will be undergone carry a 50% chance of requiring a transfusion. A technique that might lower the need for transfusions is called acute normovolemic hemodilution (ANH). ANH was first introduced over twenty years ago and has been used in many types of operations, including liver or pancreas resection. The studies done on ANH at other hospitals suggest that it may help conserve blood. Researchers at Memorial Sloan-Kettering Cancer Center are conducting a study to determine if ANH is better than the 'standard technique' that is currently used in all patients. The purpose of this study is to find out which of the two techniques is better.

The purpose of the study is to see if ANH lowers the need for the transfusion of blood products during and after liver or pancreas resection.

The second purpose of the study is to see how ANH changes the length of the operation, the length of time one spends in the hospital, and the complication rate after surgery. The researchers will also see if ANH requires any changes in the administration of anesthesia.

DETAILED DESCRIPTION:
Despite improvements in peri-operative outcome, major hepatic resection and pancreaticoduodenectomy remains associated with a high risk of major blood loss and perioperative blood transfusion.The risks associated with allogeneic blood transfusions are well-known, including immunosuppression, incompatible transfusion, and transmission of infectious agents. Clearly, efforts to reduce the use of allogeneic blood products are warranted in order to avoid potential transfusion-related complications, reduce hospital cost and avoid periods of critical blood shortage.

ANH is an approach to blood conservation that involves removal of whole blood from a patient immediately prior to an operation that is likely to be associated with significant blood loss. Following blood removal, euvolemia is restored with crystalloid and/or colloid. The harvested blood, which has a greater red cell mass than the blood lost intraoperatively, is re-infused as needed during the procedure or at the completion of the operation. ANH is more attractive than preoperative autologous blood donation for several reasons: it is technically and logistically much simpler, it requires no special equipment and costs less (no storage or administrative costs), it is associated with a lower chance of administration error, it requires no obligate pre-operative delay and is not associated with a waste of autologous units. In addition, because coagulation factors are preserved and later re-infused, ANH may reduce the need for post-operative fresh frozen plasma (FFP). Additionally, ANH may have an impact on low CVP anesthetic management during partial hepatectomy, which is standard at MSKCC and at many other centers.

The present study will help elucidate the efficacy of ANH as a means of reducing the allogeneic transfusion rate in patients undergoing major hepatic resection. If shown to be effective in reducing the use of allogeneic blood products, ANH will not only impact the current practice of hepatic resectional surgery but may also change current practice in other surgical disciplines.

This will be a prospective randomized study. Eligible patients will be consented for the trial prior to the operation.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years).
* Pre-operative hemoglobin concentration >= 11 mg/dl (males); >= 10 mg/dl (females) within 14 days of registration.
* Patients scheduled for resection of 3 or more liver segments for any indication, with or without other planned procedures or patients scheduled for pancreaticoduodenectomy

Exclusion Criteria:

* A history of active coronary artery disease. Patients with a history of coronary artery disease will be eligible if they have had a cardiac stress study showing no reversible ischemia and normal left ventricular (LV) function within 30 days of operation.
* A history of cerebrovascular disease.
* A history of congestive heart failure.
* A history of uncontrolled hypertension.
* A history of restrictive or obstructive pulmonary disease.
* A history of renal dysfunction (creatinine [Cr] > 1.8).
* Abnormal coagulation parameters (International Normalized Ratio [INR] > 1.5 not on Coumadin, or platelet count < 100,000).
* Presence of active infection.
* Evidence of hepatic metabolic disorder (bilirubin > 2 mg/dl, ALT > 75 U/L in the absence of biliary tract obstruction).
* Pre-operative autologous blood donation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 372 (Actual)
Dates: Start 2004-03; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
To determine if ANH reduces the requirement for allogeneic red cell transfusions in patients undergoing major hepatic resection or pancreaticoduodenectomy compared to standard intraoperative management | All patients will have their blood checked every 30 minutes during surgery

SECONDARY OUTCOMES:
To determine if ANH reduces the requirement for allogeneic FFP transfusions in patients undergoing major hepatic resection or pancreaticoduodenectomy compared to standard intraoperative management | All patients will have their blood checked every 30 minutes during surgery
To determine the impact of ANH on post-operative complications, length of hospital stay and operating time compared to standard intraoperative management | Two weeks
To assess the impact of ANH on low central venous pressure (CVP) anesthetic management during partial hepatectomy | Continuous monitoring during surgery

CONTACTS AND LOCATIONS:
Overall Officials: William R. Jarnagin, M.D., Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Fischer M, Matsuo K, Gonen M, Grant F, Dematteo RP, D'Angelica MI, Mascarenhas J, Brennan MF, Allen PJ, Blumgart LH, Jarnagin WR. Relationship between intraoperative fluid administration and perioperative outcome after pancreaticoduodenectomy: results of a prospective randomized trial of acute normovolemic hemodilution compared with standard intraoperative management. Ann Surg. 2010 Dec;252(6):952-8. doi: 10.1097/SLA.0b013e3181ff36b1. PMID 21107104
- [Derived] Jarnagin WR, Gonen M, Maithel SK, Fong Y, D'Angelica MI, Dematteo RP, Grant F, Wuest D, Kundu K, Blumgart LH, Fischer M. A prospective randomized trial of acute normovolemic hemodilution compared to standard intraoperative management in patients undergoing major hepatic resection. Ann Surg. 2008 Sep;248(3):360-9. doi: 10.1097/SLA.0b013e318184db08. PMID 18791356
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org